CLINICAL TRIAL: NCT06583707
Title: Effect of the Application of Real Dry Needling and Placebo Dry Needling Applied With and Without Ultrasound Guidance on the Infraspinatus Muscle in Shoulder Pain and Functionality in Patients Diagnosed With Rotator Cuff Tendinopathy
Brief Title: Real Dry Needling and Placebo Dry Needling Applied With and Without Ultrasound Guidance on the Infraspinatus Muscle
Acronym: DN-INFR-RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Enrique Coca, Student, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dry Needling Infraspinatus
Record Dates: First submitted 2024-09-01; First posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Tendinopathy; Rotator Cuff
Keywords: Dry needling; Rotator cuff; Pain; Tendinopathy; ultrasound-guided; exercise
MeSH Terms: conditions — Tendinopathy; Pain; Motor Activity | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Real ultrasound-guided dry needling on the infraspinatus muscle + exercise (Active Comparator): Patients who undergo ultrasound-guided real dry needling, using the ultrasound to visualize the needle, and who follow an exercise program.
  Interventions: Procedure: Dry needling with and without ultrasound guidance
- Placebo ultrasound-guided dry needling on the infraspinatus muscle + exercise (Sham Comparator): Patients who will undergo ultrasound-guided placebo dry needling on the infraspinatus muscle and will follow an established exercise protocol.
  Interventions: Procedure: Dry needling with and without ultrasound guidance
- Non-ultrasound-guided real dry needling on the infraspinatus muscle + exercise (Active Comparator): Patients who will undergo non-ultrasound-guided dry needling on the infraspinatus muscle and will follow an established exercise protocol
  Interventions: Procedure: Dry needling with and without ultrasound guidance
- Non-ultrasound-guided placebo dry needling on the infraspinatus muscle + exercise (Sham Comparator): Patients who will undergo non-ultrasound-guided placebo dry needling on the infraspinatus muscle and will follow an established exercise protocol
  Interventions: Procedure: Dry needling with and without ultrasound guidance

INTERVENTIONS:
Procedure: Dry needling with and without ultrasound guidance — The dry needling technique involves inserting a sterile needle to stimulate a myofascial trigger point with the aim of reducing pain and increasing range of motion and quality of life. This technique can be performed using ultrasound guidance, which allows us to visualize the needle at all times, but it can also be done using anatomical landmarks. In the placebo dry needling technique, the needle will remain stationary in the subcutaneous tissue.

SUMMARY:
The infraspinatus muscle is one of the four muscles that form the rotator cuff. The dry needling technique involves inserting a sterile needle to stimulate a myofascial trigger point with the aim of reducing pain and increasing range of motion and quality of life. This technique can be performed using ultrasound guidance, which allows us to visualize the needle at all times, but it can also be done using anatomical landmarks. This study includes a self-directed exercise plan for rotator cuff tendinopathy. Variables such as strength, shoulder functionality level, grip strength, and active range of motion will be measured. As part of the intervention, two dry needling sessions will be performed, 14 days apart, along with two different exercise programs. Three measurements will be taken, and the intervention will last for 6 weeks. The sample will be divided into four equal groups: Group 1: ultrasound-guided real dry needling; Group 2: ultrasound-guided placebo dry needling; Group 3: non-ultrasound-guided real dry needling; and Group 4: non-ultrasound-guided placebo dry needling

DETAILED DESCRIPTION:
Pathologies affecting the rotator cuff are the most common among shoulder patho-logies. The infraspinatus muscle is one of the four muscles that make up the rotator cuff. Dry needling is a technique used to reduce pain and increase the range of motion. The ul-trasound-guided technique involves using an ultrasound device to visualize the needle and guide it to the target tissue. Physical exercise helps improve tendon recovery. Objective: To evaluate the effect of real dry needling and placebo dry needling, whether ultrasound-guided or not, on pain (VAS), shoulder functionality (SPADI questionnaire), grip strength (Jamar dynamometer), and ac-tive range of motion (electronic goniometer). A total of 76 subjects diagnosed by a physician with rotator cuff tendinopathy based on imaging, aged between 18 and 60 years, and meeting the inclusion and exclusion criteria, were divided into 4 groups: Group 1 (real ultrasound-guided dry needling on the infraspinatus muscle + exercise), Group 2 (placebo ultrasound-guided dry needling on the infraspinatus muscle + exercise), Group 3 (real non-ultrasound-guided dry needling on the infraspinatus muscle + exercise), and Group 4 (placebo non-ultrasound-guided dry needling on the infraspinatus muscle + exercise). The dry needling technique will be applied twice: at the beginning and at 14 days. The intervention duration is 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

Patients aged between 18 and 60 years. Patients diagnosed with rotator cuff tendinopathy by a physician. The physician must have determined this diagnosis based on an imaging test: ultrasound or MRI. Presence of a taut band in the infraspinatus muscle with active trigger points that reproduce the patient's symptoms upon pressure.

-

Exclusion Criteria:

High-level athletes, patients diagnosed with capsulitis, patients with a history of humeral or scapular fracture, patients with a complete or partial rotator cuff tear, patients diagnosed with cancer, and patients with any contraindications related to dry needling, patients who have previously undergone shoulder surgery, patients with a history of shoulder dislocation, patients diagnosed with fibromyalgia, patients taking medication for shoulder pain, and pregnant patients

-

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-09-23 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Pain (VAS) | Before starting the treatment, at the end of the treatment, and six months after completing the treatment
  To assess the pain variable, the Visual Analog Scale (VAS) will be used. This scale consists of a range from 0 to 10, where 0 indicates no pain and 10 indicates the worst possible pain. The patient autonomously selects a number from this scale based on the level of pain they feel

SECONDARY OUTCOMES:
Shoulder functionality | Before starting the treatment, at the end of the treatment, and six months after completing the treatment
  To assess the shoulder functionality level, the Shoulder Pain and Disability Index (SPADI) questionnaire will be used. An 8-item block of questions, which addresses the disability the person feels when performing various activities, will be used to evaluate shoulder functionality. The patient will need to respond to the questions by assigning a number between 0 and 10, where 0 indicates no difficulty performing the activity and 10 represents the maximum possible difficulty in performing the activity.
Grip strength | Before starting the treatment, at the end of the treatment, and six months after completing the treatment
  To assess the grip strength variable, grip strength will be measured through an isotonic contraction using a Jamar dynamometer. Three measurements will be taken with the affected arm, asking for a contraction of 3 to 5 seconds. The highest score of the three measurements will be the final result of the test. A well-calibrated hand dynamometer must be used for this test. Kilograms (kg) will be used as the unit of measurement.
Active range of motion | Before starting the treatment, at the end of the treatment, and six months after completing the treatment
  The variable of active range of motion in the affected upper limb will be measured for flexion, abduction, internal rotation, and external rotation using a highly reliable electronic goniometer. Three measurements of each movement will be taken, and the final value will be obtained by averaging the three measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Coca, Student, Principal Investigator — University of Alcala
Locations (1):
- Campus Científico-Tecnológico UAH Av. de León, 3A, Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Serpi F, Albano D, Rapisarda S, Chianca V, Sconfienza LM, Messina C. Shoulder ultrasound: current concepts and future perspectives. J Ultrason. 2021 Jun 7;21(85):e154-e161. doi: 10.15557/JoU.2021.0025. Epub 2021 Jun 18. PMID 34258041
- [Background] de-Queiroz JHM, de-Medeiros MB, de-Lima RN, Cerdeira DQ. Exercise for rotator cuff tendinopathy. Rev Bras Med Trab. 2023 Feb 3;20(3):498-504. doi: 10.47626/1679-4435-2022-698. eCollection 2022 Jul-Sep. PMID 36793454
- [Background] Cooper K, Alexander L, Brandie D, Brown VT, Greig L, Harrison I, MacLean C, Mitchell L, Morrissey D, Moss RA, Parkinson E, Pavlova AV, Shim J, Swinton PA. Exercise therapy for tendinopathy: a mixed-methods evidence synthesis exploring feasibility, acceptability and effectiveness. Health Technol Assess. 2023 Oct;27(24):1-389. doi: 10.3310/TFWS2748. PMID 37929629
- [Background] Tahran O, Yesilyaprak SS. Effects of Modified Posterior Shoulder Stretching Exercises on Shoulder Mobility, Pain, and Dysfunction in Patients With Subacromial Impingement Syndrome. Sports Health. 2020 Mar/Apr;12(2):139-148. doi: 10.1177/1941738119900532. Epub 2020 Feb 4. PMID 32017660
- [Background] Aboelnour NH, Kamel FH, Basha MA, Azab AR, Hewidy IM, Ezzat M, Kamel NM. Combined effect of graded Thera-Band and scapular stabilization exercises on shoulder adhesive capsulitis post-mastectomy. Support Care Cancer. 2023 Mar 16;31(4):215. doi: 10.1007/s00520-023-07641-6. PMID 36922413
- [Background] Beaudart C, Rolland Y, Cruz-Jentoft AJ, Bauer JM, Sieber C, Cooper C, Al-Daghri N, Araujo de Carvalho I, Bautmans I, Bernabei R, Bruyere O, Cesari M, Cherubini A, Dawson-Hughes B, Kanis JA, Kaufman JM, Landi F, Maggi S, McCloskey E, Petermans J, Rodriguez Manas L, Reginster JY, Roller-Wirnsberger R, Schaap LA, Uebelhart D, Rizzoli R, Fielding RA. Assessment of Muscle Function and Physical Performance in Daily Clinical Practice : A position paper endorsed by the European Society for Clinical and Economic Aspects of Osteoporosis, Osteoarthritis and Musculoskeletal Diseases (ESCEO). Calcif Tissue Int. 2019 Jul;105(1):1-14. doi: 10.1007/s00223-019-00545-w. Epub 2019 Apr 10. PMID 30972475
- [Background] Wahba MM, Selim M, Hegazy MM, Elgohary R, Abdelsalam MS. Eccentric Versus Concentric Exercises in Patients With Rheumatoid Arthritis and Rotator Cuff Tendinopathy: A Randomized Comparative Study. Ann Rehabil Med. 2023 Feb;47(1):26-35. doi: 10.5535/arm.22150. Epub 2023 Feb 15. PMID 36792052
- [Background] Dupuis F, Barrett E, Dube MO, McCreesh KM, Lewis JS, Roy JS. Cryotherapy or gradual reloading exercises in acute presentations of rotator cuff tendinopathy: a randomised controlled trial. BMJ Open Sport Exerc Med. 2018 Dec 26;4(1):e000477. doi: 10.1136/bmjsem-2018-000477. eCollection 2018. PMID 30622733
- [Background] Kinsella R, Cowan SM, Watson L, Pizzari T. A comparison of isometric, isotonic concentric and isotonic eccentric exercises in the physiotherapy management of subacromial pain syndrome/rotator cuff tendinopathy: study protocol for a pilot randomised controlled trial. Pilot Feasibility Stud. 2017 Nov 14;3:45. doi: 10.1186/s40814-017-0190-3. eCollection 2017. PMID 29163981
- [Background] Roch M, Morin M, Gaudreault N. Immediate Effect of Dry Needling on the Viscoelastic Properties of a Trigger Point on the Infraspinatus Muscle Measured with MyotonPRO. Physiother Can. 2022 Jun 17;74(3):232-239. doi: 10.3138/ptc-2020-0095. eCollection 2022 Aug. PMID 37325218